CLINICAL TRIAL: NCT04893148
Title: Efficacy and Safety of iGlarLixi Versus Insulin Glargine Plus Dulaglutide in Patients With Type 2 Diabetes Insufficiently Controlled by Insulin Glargine and Metformin Combination Therapy
Brief Title: Efficacy and Safety of iGlarLixi Versus Insulin Glargine Plus Dulaglutide in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chungbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Eu Jeong Ku, Clinical Associate Professor, Chungbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLP1RA2021
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Type 2 Diabetes Mellitus; Glucose, High Blood
Keywords: IGlarLixi; Dulaglutide; Continuous glucose monitoring system; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iGlar/Lixi (Active Comparator): Switching to IGlarLixi from insulin glargine iGlar/Lixi starts with the following doses depending on the existing insulin glargine dose: 1) insulin glargine <20 unit/day = iGlar/Lixi 10 unit/day, 2) insulin glargine >=20 unit/day = iGlar/Lixi 20 unit/day.
  Training to increase the iGlar/Lixi dosage every 3 days to meet the target fasting blood glucose level to 80~130 mg/day
  Interventions: Drug: IGlarLixi
- Dulaglutide plus insulin glargine (Active Comparator): Adding Dulaglutide to insulin glargine. Keep insulin glargine and dulaglutide start at 0.75 mg per week and increase to 1.5 mg per week after 1 month with evaluating compliance and tolerability.
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: IGlarLixi — Changing to iGlarLixi from insulin glargine
  Arms: iGlar/Lixi
Drug: Dulaglutide — Add dulaglutide to insulin glargine
  Other Names: Insulin Glargine
  Arms: Dulaglutide plus insulin glargine

SUMMARY:
The investigators aimed to compare efficacy and safety of IGlarLixi and insulin glargine plus dulaglutide as intensification from basal insulin with metformin, in the absence of head-to-head trials.

DETAILED DESCRIPTION:
Fixed-dose combinations of insulin glargine/lixisenatide (IGlarLixi) or insulin glargine plus dulaglutide constitute treatment intensification in type 2 diabetes mellitus (T2D). The investigators aimed to compare efficacy and safety of IGlarLixi and insulin glargine plus dulaglutide as intensification from basal insulin with metformin, in the absence of head-to-head trials. Treatments were compared in terms of glycated hemoglobin (HbA1c), fasting plasma glucose (FPG) change from baseline, and variables from continuous glucose monitoring (CGM) system; in addition to safety issues on hypoglycemia and changes in weight.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient with type 2 diabetes, treated with basal insulin plus metformin (maximum tolerated dosage) for at least 12 weeks
* Patient accepting to participant to this study

Exclusion Criteria:

* Pregnant or breastfeeding woman
* severe renal dysfunction (eGFR <60 ml/min/1.73m2)
* chronic or acute hepatic disorder (HBV or HCV hepatitis, liver cirrhosis etc.) (AST/ALT > 2.5*ULN)
* Prescription such as immunosuppressant agents, glucocorticoids
* Active anti-cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in glycated hemoglobin (HbA1c) | Baseline, week 12
  HbA1c will be measured at baseline and week 12

SECONDARY OUTCOMES:
Changes in fasting plasma glucose (FPG) | Baseline, week 12
  Comparison of FPG changes in week 12 from baseline between the two groups
Changes in glucose time in range (TIR) | Baseline, week 12
  Comparison of %TIR changes in week 12 from baseline between the two groups
Changes in glucose time above range (TAR) | Baseline, week 12
  Comparison of %TAR changes in week 12 from baseline between the two groups
Changes in glucose time below range (TBR) | Baseline, week 12
  Comparison of %TBR changes in week 12 from baseline between the two groups
Incidence of hypoglycemia | Baseline, week 12
  Comparison of the incidence of hypoglycemia between the two groups
Changes in weight | Baseline, week 12
  Comparison of weight changes in week 12 from baseline between the two

CONTACTS AND LOCATIONS:
Overall Officials: Eu Jeong Ku, MD, PhD, Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Chungbuk National University Hospital, Cheonju, North Chungcheong, South Korea